CLINICAL TRIAL: NCT01502696
Title: Adjuvant Pegylated-Interferon-alpha2b (SylatronTM) for 2 Years Versus Observation in Patients With an Ulcerated Primary Cutaneous Melanoma With T(2-4)bN0M0: a Randomized Phase III Trial of the EORTC Melanoma Group.
Brief Title: Adjuvant PEG Intron in Ulcerated Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-18081; 2009-010273-20 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2012-01-02 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Ulcerated Melanomas
Keywords: ulcerated primary cutaneous melanoma; Stage II; PEG IFN alfa-2b; T(2-4)bN0M0
MeSH Terms: interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG IFN alfa-2b (Experimental)
  Interventions: Biological: PEG IFN alfa-2b
- Observation (No Intervention)

INTERVENTIONS:
Biological: PEG IFN alfa-2b — 3µg/kg weekly injections
  Arms: PEG IFN alfa-2b

SUMMARY:
Patients with an ulcerated melanoma with Breslow >1 mm, N0M0 have a significantly higher risk for relapse than patients with a non-ulcerated primary and about a 40-50% chance of developing stage IV disease to which they will almost invariably succumb. In stage I and II patients with an ulcerated primary who have been sentinel node (SN-staged) and found to be SN-negative there is still a 25-30% relapse risk.

The purpose of this study is to evaluate the effectiveness and safety when treated with PEG IFN alfa-2b for 2 years as compared to observation (no treatment), administered after adequate surgery has been performed for ulcerated primary cutaneous melanomas.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18-70 years old.
* Subjects must have histologically documented ulcerated primary cutaneous melanomas with T(2-4)b N0M0.

Adequate resection of ulcerated primary cutaneous melanoma. 1 to 2 cm normal tissue excision margins according to Breslow thickness are recommended. In the head and neck areas and in case of locations distally on extremities, narrower margins are acceptable as long as they are radical (see Appendix F). Subjects must have recovered from the effects of recent surgery.

* SNB must occur within 12 weeks prior randomization.
* Subjects must have an ECOG performance status of 0 or 1 (See Appendix B).
* Subjects must have adequate bone marrow, renal and hepatic function as defined by the following parameters obtained up to maximum 12 weeks prior to randomization:

  * Hematology:
  * WBC >= 3.0 x 109/L
  * Neutrophils > 1.5 x 109/L
  * Platelets > 100 x 109/L
  * Hemoglobin >= 9 g/dL or 5.6 mmol/L
  * Adequate Renal and Hepatic function:
  * Serum creatinine < 2.0 mg/dL or < 140 µmol/L
  * SGOT and SGPT < 2 times upper normal limit of laboratory normal (ULN)

Exclusion Criteria:

* No mucosal melanoma nor ocular melanoma.
* No evidence of nodal involvement confirmed by sentinel lymph node biopsy (SNB). Sentinel Node staging after the excision of the primary must be done between the date of final excision of the primary and the date of randomization.
* No evidence of regional nor distant lymph node metastases nor satellites/in-transit metastases (even if they have been resected).
* No evidence of distant metastasis on clinical examination, CT/MRI of full chest, abdomen and pelvis. Neck CT/MRI if head and neck primary.
* No clinical evidence of brain metastasis.
* No pregnant women
* No breast feeding women
* No patients with a medical condition requiring chronic systemic corticosteroids are not eligible.
* No experimental therapy within 30 days prior to randomization in this study.
* No prior chemotherapy, immunotherapy/vaccine, hormonal or radiation therapy for melanoma.
* No prior treatment with interferon-alfa for any reason.
* No history of prior malignancy within the past 5 years other than surgically cured non-melanoma skin cancer or cervical carcinoma in situ.
* No severe cardiovascular disease, i.e. arrhythmias requiring chronic treatment, congestive heart failure (NYHA Class III or IV) nor symptomatic ischemic heart disease.
* No thyroid dysfunction not responsive to therapy.
* No poorly controlled (HBA1C>8%) diabetes mellitus or uncontrolled diabetes mellitus, i.e. elevated fasting serum glucose should be < 110% ULN).
* No active autoimmune disease.
* No active and/or uncontrolled infection, including active hepatitis.
* No history of seropositivity for HIV.
* No history of neuropsychiatric disorder requiring hospitalization.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2012-10; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 6.3 years from first patient in

SECONDARY OUTCOMES:
Occurence of Adverse Events | 6.3 years from first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.
Overall survival (OS) | 7.8 years from first patient in
Distant metastases-free survival (DMFS) | 7.8 years from first patient in
Quality of life | 6 years from from first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Eggermont, MD, PHD, Study Chair — Institut Gustave Roussy, Paris, France
Locations (57):
- Medical University of Graz, Graz, Austria
- Belgium (3):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital - University Copenhagen, Herlev
  - Odense University Hospital, Odense
- France (14):
  - Assistance Publique - Hopitaux de Paris - Hopital Avicenne, Bobigny
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre (Bordeaux, France, Bordeaux
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - CHRU de Lille, Lille
  - Centre Leon Berard, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone, Marseille
  - CHU de Nice - CHU de Nice - Hopital De L'Archet, Nice
  - Assistance Publique - Hopitaux de Paris - CHU Ambroise Pare, Paris
  - Assitance Publique - Hopitaux de Paris - Hopital Bichat-Claude Bernard, Paris
  - Assitance Publique - Hopitaux de Paris - Hopital Saint-Louis, Paris
  - Institut Gustave Roussy, Paris
  - Centre Hospitalier De Pau, Pau
  - CHU de Reims - Hôpital Robert Debré, Reims
  - CHU d'Amiens - CHU Amiens - Hopital Sud, Salouël
- Germany (9):
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum, Essen
  - Universitaetsklinikum Heidelberg - Hautklinik / Dermatologic Department, Heidelberg
  - Universitaetsklinikum Heidelberg - Hautklinik, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Medizinische Universitaet Zu Luebeck, Lübeck
  - Johannes Gutenberg Universitaetskliniken - Mainz University Medical Center, Mainz
  - UniversitaetsMedizin Mannheim, Mannheim
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (5):
  - IRCCS - Istituto Tumori "Giovanni Paolo II", Bari
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Istituto Dermopatico Dell'Immacolata, Roma
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia" di Udine, Udine
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Leiden University Medical Centre, Leiden
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Portugal (2):
  - I.P.O. Francisco Gentil - Centro De Lisboa, Lisbon
  - Hospital Distrital De Santarem, Santarém
- Spain (2):
  - Hospital Clinic Universitari, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- UniversitaetsSpital Zurich, Zurich, Switzerland
- United Kingdom (13):
  - Clatterbridge Centre for Oncology NHS Trust - Clatterbridge Cancer Centre NHS Foundation Trust, Bebington
  - University Hospitals Birmingham NHS Foundation Trust (UHB) - Queen Elisabeth Medical Centre, Birmingham
  - Mid Essex Hospitals - Broomfield Hospital, Broomfield
  - Cambridge University Hospital NHS - Addenbrookes Hospital, Cambridge
  - Cheltenham General Hospital, Cheltenham
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - St George's Hospital NHS Trust (6961), London
  - The Christie NHS Foundation Trust, Manchester
  - Norfolk And Norwich Hospital, Norwich
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton
  - St Helens and Knowsley Teaching Hospitals, St Helens